CLINICAL TRIAL: NCT02985814
Title: Identifying Patients With the COPD-Asthma Overlap Phenotype: Therapeutic Implications
Status: Completed | Type: Observational
Sponsor: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 0066-14-COM
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: COPD Asthma
Keywords: COPD Asthma Overlap

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with airway obstruction: Patients referred for pulmonary function test diagnosed with airway obstruction (FEV1/FVC < 0.7) willing to sign an informed consent.

SUMMARY:
Background: Asthma and COPD are considered different diseases but many patients share characteristics of both entities. This has been termed "COPD-asthma overlap syndrome".

Study objective: To examine: (a) the frequency of the overlap phenotype among patients referred for pulmonary function testing and, (b) the impact of this phenotype on the therapeutic management and the quality of life of these patients as compared with patients with COPD only and asthma only.

Methods:

Type of study: Observational, cross-sectional. Study subjects: Patients referred for pulmonary function test diagnosed with airway obstruction (FEV1/FVC < 0.7) willing to sign an informed consent.

Study procedures: Spirometry will be performed before and after the administration of a bronchodilator. Respiratory questionnaire: Questionnaires about smoking habits, past history of asthma and wheezing, current medications and history of exacerbations will be administered at inclusion. Questionnaire on medication utilization will be administered by telephone one month after inclusion. Quality of life: Will be assessed using the Saint George Respiratory Questionnaire (SGRQ).

Working definitions: The following definitions will be adopted: a) COPD only: smoking history > 10 pack/years and post-bronchodilator (BD) FEV1/FVC ratio of < 0.70; b) Asthma only: (1) presence of wheezing in the last year plus a minimum post-BD increase in FEV1 or FVC of 12% and 200 ml; (2) prior physician diagnosis (before age 40); and c) both COPD-Asthma (the overlap group) - the combination of the two.

Outcome measures: The clinical outcome is the prevalence rate of the phenotypes. Patient-reported outcomes will include the utilization of medication, the number of exacerbations, and quality of life.

DETAILED DESCRIPTION:
Background: Asthma and COPD are considered different diseases but many patients share characteristics of both entities. This has been termed "COPD-asthma overlap syndrome".

Study objective: To examine: (a) the frequency of the overlap phenotype among patients referred for pulmonary function testing and, (b) the impact of this phenotype on the therapeutic management and the quality of life of these patients as compared with patients with COPD only and asthma only.

Methods:

Type of study: Observational, cross-sectional. Study subjects: Patients referred for pulmonary function test diagnosed with airway obstruction (FEV1/FVC < 0.7) willing to sign an informed consent.

Study procedures: Spirometry will be performed before and after the administration of a bronchodilator. Respiratory questionnaire: Questionnaires about smoking habits, past history of asthma and wheezing, current medications and history of exacerbations will be administered at inclusion. Questionnaire on medication utilization will be administered by telephone one month after inclusion. Quality of life: Will be assessed using the Saint George Respiratory Questionnaire (SGRQ).

Working definitions: The following definitions will be adopted: a) COPD only: smoking history > 10 pack/years and post-bronchodilator (BD) FEV1/FVC ratio of < 0.70; b) Asthma only: (1) presence of wheezing in the last year plus a minimum post-BD increase in FEV1 or FVC of 12% and 200 ml; (2) prior physician diagnosis (before age 40); and c) both COPD-Asthma (the overlap group) - the combination of the two.

Outcome measures: The clinical outcome is the prevalence rate of the phenotypes. Patient-reported outcomes will include the utilization of medication, the number of exacerbations, and quality of life.

Statistical plan: Sample size: For an estimated prevalence rate of 20%, 246 patients should be recruited with 5% imprecision and 95% degree of confidence. To round up, 250 patients will be included. Statistical methods: Multiple comparisons will be carried out using the one-way ANOVA for continuous variables and chi-squared test (or Fisher Exact Test) for qualitative variables. Multiple logistic regression models will be tested to examine the relation between the "COPD-asthma overlap" phenotype and various independent or predictor variables.

Expected benefits: Data collected could serve to advance the medical community's knowledge pertaining to the COPD-asthma overlap syndrome. Most importantly, however, they will encourage reflection on the best therapeutic options for the patients with the overlap syndrome. Indeed, recommendations on this matter are noticeably absent from the current guidelines proposed to treat and monitor obstructive lung diseases.

ELIGIBILITY:
Inclusion Criteria:

men or women aged > 18 years , with spirometric evidence of airway obstruction defined as an FEV1/FVC ratio < 0.7

Exclusion Criteria:

Subjects with normal spirometry or presenting a pattern of restrictive lung disease will be listed for the purpose of characterising the source population but will not enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men or women aged > 18 years, with spirometric evidence of airway obstruction defined as an FEV1/FVC ratio < 0.7
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
utilization of medication | enrollment to 2 months
  completion of RS questionnaires

SECONDARY OUTCOMES:
number of exacerbations | enrollment to 2 months
  completion of RS questionnaires
quality of life | enrollment
  completion of Saint George Respiratory Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel IZBICKI, MD, Principal Investigator — Clalit Health Services
Locations (1):
- ROKACH institute, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No